CLINICAL TRIAL: NCT05751330
Title: Efficacy of Transcatheter Ablation of Ganglionic Plexuses (Cardioneuroablation) in Right Atrium in Patients With Asystolic Neuromediated Syncope
Brief Title: Italian Cardioneuroablation Study for Neurocardiogenic Syncope Patients
Acronym: ItalianCNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Casilino ASL RMB (Other)
Collaborators: Gruppo Italiano Multidisciplinare per lo Studio della Sincope (Other)
Responsible Party: Principal Investigator, Leonardo Calò, MD, Professor, Policlinico Casilino ASL RMB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCasilino
Record Dates: First submitted 2023-01-04; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Neurally Mediated Syncope
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients affected by Cardioinhibitory Neurocardiogenic Syncope (Experimental)
  Interventions: Procedure: Transcatheter ablation of cardiac ganglionated plexi

INTERVENTIONS:
Procedure: Transcatheter ablation of cardiac ganglionated plexi — The ablative procedure involves applying radiofrequency deliveries in the two
  Right atrium anatomical sites close to the two main ganglionic plexuses of the right atrium:
  * Inferior-posterior area (site of first ablation) corresponding to the right inferior atrial ganglion located between the inferior vena cava, coronary sinus ostium and near the atrioventricular node
  * Upper-posterior area (site of second ablation) corresponding to the right superior atrial ganglion located between the superior vena cava and the posterior surface of the right atrium

SUMMARY:
Multicenter Italian interventional "proof of efficacy" clinical trial that aims to evaluate the incidence of asystolic pauses and heart rate in patients with CNS who performed severe CNA identified through asystolic pauses identification by implantable loop recorder. The study is independent, "investigator-initiated," sponsored by a nonprofit scientific association called the Italian Multidisciplinary Group for the Study of Syncope (GIMSI).

DETAILED DESCRIPTION:
The so called "Cardioneuroablation (CNA)" focused on the endocardial ablation of atrial ganglionated plexi has proven to be efficacy in patients affected by neuro-mediated cardioinhibitory syncope (NCS). No center currently has sufficient case series to establish long-term efficacy and safety results, for which a multicenter interventional study is therefore needed.

The aim of the study will be to evaluate the efficacy and safety of CNA focused in NCS patients. The ablation procedure, consists of radiofrequency delivering at right atrial anatomic sites where the underlying presence of GP clusters is regarded as highly probable: 1) the inferior-posterior area (first ablation site): inferior right GP placed between inferior vena cava, coronary sinus ostium and near the atrio-ventricular groove, 2) the superior-posterior area (second ablation site): superior right atrial GP, adjacent to the junction of the superior vena cava and the posterior surface of RA.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Patients with a clinical diagnosis of neuromediated syncope according to class I criteria of the ESC guidelines, Table 1
* Clinical history of recurrent syncope (≥2 in the last year or ≥3 in the last 2 years), severe, not tolerated by the patient
* Documentation of ≥2 asystolic pauses >3 sec daytime on ECG monitoring by implantable loop recorder (ILR), with or without syncope
* Refusal by patient to perform pacemaker implantation

Tilt test is recommended but not mandatory. Patients with negative tilt test are also enrollable. It can be either positive or negative.

Exclusion Criteria:

* Absence of sinus dysfunction and atrioventricular node disease.
* Absence of structural heart disease
* Possible alternative diagnoses of syncope

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Intrapatient incidence of asystolic episodes before and after cardioneuroablation | through study completion, an average of 1 year
  frequency (number and percentage) of asystolic episodes before and after ablation

SECONDARY OUTCOMES:
Comparison of mean heart rate, before and after cardioneuroablation, incidence of (pre)syncopal episodes before and after CNA and, finally, beat-to beat HR variability during ILR monitoring | through study completion, an average of 1 year
  intrapatient comparison of mean heart rate (bpm), beat-to-beat variability of heart rate, before and after CNA.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Casilino, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Yes
The study envisages the subsequent activation of other participating centres to recruit and enrol patients to undergo the Cardioneuroablation procedure
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Task Force for the Diagnosis and Management of Syncope; European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Heart Failure Association (HFA); Heart Rhythm Society (HRS); Moya A, Sutton R, Ammirati F, Blanc JJ, Brignole M, Dahm JB, Deharo JC, Gajek J, Gjesdal K, Krahn A, Massin M, Pepi M, Pezawas T, Ruiz Granell R, Sarasin F, Ungar A, van Dijk JG, Walma EP, Wieling W. Guidelines for the diagnosis and management of syncope (version 2009). Eur Heart J. 2009 Nov;30(21):2631-71. doi: 10.1093/eurheartj/ehp298. Epub 2009 Aug 27. No abstract available. PMID 19713422
- [Result] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Result] Sutton R, Petersen ME. The clinical spectrum of neurocardiogenic syncope. J Cardiovasc Electrophysiol. 1995 Jul;6(7):569-76. doi: 10.1111/j.1540-8167.1995.tb00429.x. PMID 8528491
- [Result] Brignole M, Menozzi C, Moya A, Andresen D, Blanc JJ, Krahn AD, Wieling W, Beiras X, Deharo JC, Russo V, Tomaino M, Sutton R; International Study on Syncope of Uncertain Etiology 3 (ISSUE-3) Investigators. Pacemaker therapy in patients with neurally mediated syncope and documented asystole: Third International Study on Syncope of Uncertain Etiology (ISSUE-3): a randomized trial. Circulation. 2012 May 29;125(21):2566-71. doi: 10.1161/CIRCULATIONAHA.111.082313. Epub 2012 May 7. PMID 22565936
- [Result] Soteriades ES, Evans JC, Larson MG, Chen MH, Chen L, Benjamin EJ, Levy D. Incidence and prognosis of syncope. N Engl J Med. 2002 Sep 19;347(12):878-85. doi: 10.1056/NEJMoa012407. PMID 12239256
- [Result] Brignole M, Russo V, Arabia F, Oliveira M, Pedrote A, Aerts A, Rapacciuolo A, Boveda S, Deharo JC, Maglia G, Nigro G, Giacopelli D, Gargaro A, Tomaino M; BioSync CLS trial Investigators. Cardiac pacing in severe recurrent reflex syncope and tilt-induced asystole. Eur Heart J. 2021 Feb 1;42(5):508-516. doi: 10.1093/eurheartj/ehaa936. PMID 33279955
- [Result] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Result] Scanavacca M, Hachul D, Pisani C, Sosa E. Selective vagal denervation of the sinus and atrioventricular nodes, guided by vagal reflexes induced by high frequency stimulation, to treat refractory neurally mediated syncope. J Cardiovasc Electrophysiol. 2009 May;20(5):558-63. doi: 10.1111/j.1540-8167.2008.01385.x. Epub 2008 Dec 17. PMID 19207753
- [Result] Armour JA, Murphy DA, Yuan BX, Macdonald S, Hopkins DA. Gross and microscopic anatomy of the human intrinsic cardiac nervous system. Anat Rec. 1997 Feb;247(2):289-98. doi: 10.1002/(SICI)1097-0185(199702)247:23.0.CO;2-L. PMID 9026008
- [Result] Singh S, Johnson PI, Lee RE, Orfei E, Lonchyna VA, Sullivan HJ, Montoya A, Tran H, Wehrmacher WH, Wurster RD. Topography of cardiac ganglia in the adult human heart. J Thorac Cardiovasc Surg. 1996 Oct;112(4):943-53. doi: 10.1016/S0022-5223(96)70094-6. PMID 8873720
- [Result] Chiou CW, Eble JN, Zipes DP. Efferent vagal innervation of the canine atria and sinus and atrioventricular nodes. The third fat pad. Circulation. 1997 Jun 3;95(11):2573-84. doi: 10.1161/01.cir.95.11.2573. PMID 9184589
- [Result] Po SS, Nakagawa H, Jackman WM. Localization of left atrial ganglionated plexi in patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2009 Oct;20(10):1186-9. doi: 10.1111/j.1540-8167.2009.01515.x. Epub 2009 Jun 26. PMID 19563367
- [Result] Calo L, Rebecchi M, Sette A, Sciarra L, Borrelli A, Scara A, Grieco D, Politano A, Sgueglia M, De Luca L, Martino A, Panattoni G, Golia P, Turrisi OV, Knowles M, Strano S, de Ruvo E. Catheter ablation of right atrial ganglionated plexi to treat cardioinhibitory neurocardiogenic syncope: a long-term follow-up prospective study. J Interv Card Electrophysiol. 2021 Sep;61(3):499-510. doi: 10.1007/s10840-020-00840-9. Epub 2020 Aug 6. PMID 32766945
- [Result] Rebecchi M, de Ruvo E, Strano S, Sciarra L, Golia P, Martino A, Calo L. Ganglionated plexi ablation in right atrium to treat cardioinhibitory neurocardiogenic syncope. J Interv Card Electrophysiol. 2012 Sep;34(3):231-5. doi: 10.1007/s10840-012-9666-5. Epub 2012 Mar 21. No abstract available. PMID 22434334
- [Result] Debruyne P, Rossenbacker T, Collienne C, Roosen J, Ector B, Janssens L, Charlier F, Vankelecom B, Dewilde W, Wijns W. Unifocal Right-Sided Ablation Treatment for Neurally Mediated Syncope and Functional Sinus Node Dysfunction Under Computed Tomographic Guidance. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006604. doi: 10.1161/CIRCEP.118.006604. PMID 30354289
- [Result] Brignole M, Iori M, Solari D, Bottoni N, Rivasi G, Ungar A, Deharo JC, Guieu R. Efficacy of theophylline in patients with syncope without prodromes with normal heart and normal ECG. Int J Cardiol. 2019 Aug 15;289:70-73. doi: 10.1016/j.ijcard.2019.03.043. Epub 2019 Mar 22. PMID 30928258

DOCUMENTS (1):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT05751330/Prot_000.pdf